CLINICAL TRIAL: NCT02566200
Title: French Registry of Acute ST-elevation or Non-ST-elevation Myocardial Infarction 2015
Acronym: FASTMI2015
Status: Active, not recruiting | Type: Observational
Sponsor: French Cardiology Society (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 15597
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Myocardial Infarction
Keywords: Acute coronary syndrome; Cardiology
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — * blood samples for genotyping and serum banking
  * faeces samples for genetic analysis of microbiota
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IM group: Patients admitted in intensive care for a myocardial infarction

SUMMARY:
Over the last two decades, considerable progress has been made in the management of myocardial infarction, both in the acute phase and in monitoring beyond the hospital phase. However changing practices in the "real world" and their impact on prognosis in the medium and long term patients admitted to the intensive care unit for acute myocardial infarction are relatively little studied exhaustively.

The study of clinical, biological and genetic characteristics of patients and their conditions of care, help to identify patients at risk for increased morbidity and mortality after myocardial infarction and could be the basis for the subsequent realization of specific studies on the optimal therapeutic management of the disease according to the different risk profiles.

DETAILED DESCRIPTION:
This is a multicenter observational study, given to 300 prospective medical facilities, including a clinic or intensive care unit entitled to receive emergency acute coronary syndromes.

Patients will be recruited consecutively during a period of 2 months.

Annual follow-ups will be conducted during 10 years of clinical research technicians of the French Society of Cardiology, mail and / or telephone contact with the municipalities of birth, treating physicians and patients.

The ambition of the 2015 Observatory of the French Society of Cardiology is through a photograph "scale" of the practices in France at present, to ensure consistency in the quality of care for hospitalized patients heart attack; the investigation will emphasize the strengths but also the weaknesses of our health care system so that should improve. Finally, the observation of a large population of the real world will give the opportunity to assess the interactions between the different types of treatments used and check their possible synergy or incompatibilities.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged over 18 years
2. Patients admitted within 48 hours of onset of symptoms in a coronary intensive care unit (USIC) for acute myocardial infarction (MI) defined by:

   A rise and fall of typical troponin (or CPKMb) associated with at least one of the following:
   * symptoms consistent with myocardial ischemia
   * development of pathological Q waves
   * repolarisation disorders related to ischemia (or in addition to ST depression, T wave inversion)
3. And having agreed to participate in the study.

Exclusion Criteria:

1. Refusal to consent
2. MI occurring in the 48 hours after therapeutic intervention (bypass surgery or coronary angioplasty or other surgical procedure)
3. Diagnosis of myocardial reversed in favor of an alternative diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient hospitalized in an intensive care unit in France for an acute myocardial infarction
Sampling Method: Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
All cause mortality 1 year after hospitalization for a myocardial infarction | 1 year after hospitalization

SECONDARY OUTCOMES:
All cause mortality 10 years after hospitalization for a myocardial infarction | 10 years after hospitalization
To determine the impact of genetic, serology, fecal biomarkers on the myocardial infarction and its complications. | 10 years after hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Danchin, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- HEGP, Paris, France

REFERENCES:
- [Result] Puymirat E, Simon T, Cayla G, Cottin Y, Elbaz M, Coste P, Lemesle G, Motreff P, Popovic B, Khalife K, Labeque JN, Perret T, Le Ray C, Orion L, Jouve B, Blanchard D, Peycher P, Silvain J, Steg PG, Goldstein P, Gueret P, Belle L, Aissaoui N, Ferrieres J, Schiele F, Danchin N; USIK, USIC 2000, and FAST-MI investigators. Acute Myocardial Infarction: Changes in Patient Characteristics, Management, and 6-Month Outcomes Over a Period of 20 Years in the FAST-MI Program (French Registry of Acute ST-Elevation or Non-ST-Elevation Myocardial Infarction) 1995 to 2015. Circulation. 2017 Nov 14;136(20):1908-1919. doi: 10.1161/CIRCULATIONAHA.117.030798. Epub 2017 Aug 27. PMID 28844989
- [Result] Belle L, Cayla G, Cottin Y, Coste P, Khalife K, Labeque JN, Farah B, Perret T, Goldstein P, Gueugniaud PY, Braun F, Gauthier J, Gilard M, Le Heuzey JY, Naccache N, Drouet E, Bataille V, Ferrieres J, Puymirat E, Schiele F, Simon T, Danchin N; FAST-MI 2015 investigators. French Registry on Acute ST-elevation and non-ST-elevation Myocardial Infarction 2015 (FAST-MI 2015). Design and baseline data. Arch Cardiovasc Dis. 2017 Jun-Jul;110(6-7):366-378. doi: 10.1016/j.acvd.2017.05.001. Epub 2017 Jun 21. PMID 28647465
- [Result] Puymirat E, Simon T, Danchin N; FAST-MI Investigators. Response by Puymirat et al to Letter Regarding Article, "Acute Myocardial Infarction Changes in Patient Characteristics, Management, and 6-Month Outcomes Over a Period of 20 Years in the FAST-MI Program (French Registry of Acute ST Elevation or Non-ST-Elevation Myocardial Infarction) 1995 to 2015". Circulation. 2018 May 22;137(21):2307-2308. doi: 10.1161/CIRCULATIONAHA.118.033969. No abstract available. PMID 29784688
- [Result] Puymirat E, Cayla G, Cottin Y, Elbaz M, Henry P, Gerbaud E, Lemesle G, Popovic B, Labeque JN, Roubille F, Andrieu S, Farah B, Schiele F, Ferrieres J, Simon T, Danchin N. Twenty-year trends in profile, management and outcomes of patients with ST-segment elevation myocardial infarction according to use of reperfusion therapy: Data from the FAST-MI program 1995-2015. Am Heart J. 2019 Aug;214:97-106. doi: 10.1016/j.ahj.2019.05.007. Epub 2019 May 16. PMID 31181374
- [Result] Puymirat E, Bonaca M, Iliou MC, Tea V, Ducrocq G, Douard H, Labrunee M, Plastaras P, Chevallereau P, Taldir G, Bataille V, Ferrieres J, Schiele F, Simon T, Danchin N; FAST-MI investigators. Outcome associated with prescription of cardiac rehabilitation according to predicted risk after acute myocardial infarction: Insights from the FAST-MI registries. Arch Cardiovasc Dis. 2019 Aug-Sep;112(8-9):459-468. doi: 10.1016/j.acvd.2019.04.002. Epub 2019 May 22. PMID 31126738
- [Result] Schiele F, Puymirat E, Ferrieres J, Simon T, Fox KAA, Eikelboom J, Danchin N; FAST-MI investigators. The FAST-MI 2005-2010-2015 registries in the light of the COMPASS trial: The COMPASS criteria applied to a post-MI population. Int J Cardiol. 2019 Mar 1;278:7-13. doi: 10.1016/j.ijcard.2018.11.138. Epub 2018 Dec 3. PMID 30538057
- [Result] Puymirat E, Bonaca M, Fumery M, Tea V, Aissaoui N, Lemesles G, Bonello L, Ducrocq G, Cayla G, Ferrieres J, Schiele F, Simon T, Danchin N; FAST-MI investigators. Atherothrombotic risk stratification after acute myocardial infarction: The Thrombolysis in Myocardial Infarction Risk Score for Secondary Prevention in the light of the French Registry of Acute ST Elevation or non-ST Elevation Myocardial Infarction registries. Clin Cardiol. 2019 Feb;42(2):227-234. doi: 10.1002/clc.23131. Epub 2018 Dec 27. PMID 30536449
- [Derived] Fayol A, Schiele F, Ferrieres J, Puymirat E, Bataille V, Tea V, Chamandi C, Albert F, Lemesle G, Cayla G, Weizman O, Simon T, Danchin N; FAST-MI Investigators. Association of Use and Dose of Lipid-Lowering Therapy Post Acute Myocardial Infarction With 5-Year Survival in Older Adults. Circ Cardiovasc Qual Outcomes. 2024 May;17(5):e010685. doi: 10.1161/CIRCOUTCOMES.123.010685. Epub 2024 Apr 29. PMID 38682335
- [Derived] Garcia R, Marijon E, Karam N, Narayanan K, Anselme F, Cesari O, Champ-Rigot L, Manenti V, Martins R, Puymirat E, Ferrieres J, Schiele F, Simon T, Danchin N. Ventricular fibrillation in acute myocardial infarction: 20-year trends in the FAST-MI study. Eur Heart J. 2022 Dec 14;43(47):4887-4896. doi: 10.1093/eurheartj/ehac579. PMID 36303402
- [Derived] Danchin N, Puymirat E, Cayla G, Cottin Y, Coste P, Gilard M, Goldstein P, Braun F, Belle L, Montalescot G, Ferrieres J, Schiele F, Simon T; FAST-MI Investigators. One-Year Survival After ST-Segment-Elevation Myocardial Infarction in Relation With Prehospital Administration of Dual Antiplatelet Therapy. Circ Cardiovasc Interv. 2018 Sep;11(9):e007241. doi: 10.1161/CIRCINTERVENTIONS.118.007241. PMID 30354592